CLINICAL TRIAL: NCT00542750
Title: An Open-Label Trial of N-Acetylcysteine in Cannabis Dependent Adolescents
Acronym: NAC MJ Pilot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Kevin Gray, MD, Professor of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5K12 DA 000357 NAC MJ Pilot; K12DA000357 (NIH)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Cannabis Dependence
Keywords: Cannabis; Marijuana; Pharmacotherapy; Adolescent
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-Acetylcysteine (Experimental): All participants will receive N-Acetylcysteine 1200 mg twice daily during four weeks of participation. Tolerability, marijuana use, and reactivity to marijuana cues will be investigated.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine 1200 mg twice daily for four weeks
  Other Names: GNC brand USP-grade NAC (600 mg capsules)

SUMMARY:
The purpose of this pilot study is to determine the feasibility of conducting a trial of N-Acetylcysteine in cannabis dependent adolescents.

DETAILED DESCRIPTION:
This project involves investigation of oral N-acetylcysteine (NAC) as a potential pharmacologic agent for treatment of cannabis dependence in adolescents. Cannabis dependence continues to be a major problem among adolescents in the United States. To date, psychosocial interventions have produced only small to modest effect sizes in controlled trials, and minimal work has been done to investigate the potential role for pharmacotherapy for cannabis dependence. Translating preclinical research suggesting a role for NAC in cocaine dependent individuals, our research group has developed preliminary evidence of decreased cocaine use and cue reactivity in humans taking NAC. Preclinical research has additionally demonstrated significant parallels in glutamatergic dysfunction in the nucleus accumbens (the proposed target of NAC treatment) between habitual cocaine and marijuana users. NAC is an inexpensive, long-available agent with a favorable tolerability profile in adults and children. However, it has not yet been studied in cannabis dependent adolescents. Hence, we are undertaking an open-label pilot trial of NAC in adolescents with cannabis dependence.

The primary specific aims of the proposed project are:

1. To assess the feasibility of conducting a trial of NAC in cannabis dependent adolescents.
2. To assess the safety and tolerability of NAC in cannabis dependent adolescents

   The secondary specific aim of the proposed project is:
3. To gather variability information to assist in design of a larger-scale, adequately powered clinical trial of NAC in cannabis dependent adolescents.

Primary hypotheses

1. It will be feasible to recruit and retain cannabis dependent adolescents in a trial of NAC.
2. NAC will be well tolerated among cannabis dependent adolescents.

   Secondary hypothesis
3. Adequate variability information will be gathered to design a larger-scale, adequately powered clinical trial of NAC in cannabis dependent adolescents.

Twenty-four adolescents between 12 and 20 years old will be recruited in this study. Results from this project will be used to design further studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 - 20 years old.
* Participants must be regular smokers of marijuana (on average smoke at least 3 times per week for at least one year) and meet DSM-IV Criteria for cannabis dependence, with desire to cut down on marijuana use.
* Participants must understand all oral and written informed consent and give such consent prior to on-site screening.
* Participants must agree to refrain from marijuana use for 24 hours prior to each cue reactivity session (Visits 2 and 4).
* Participants must have a person that can be contacted in case of emergency.
* Participants must have had stable residence for the past 30 days.
* Post-menarchal female participants must agree to use birth control to avoid pregnancy.

Exclusion Criteria:

* Allergy or intolerance to N-Acetylcysteine (NAC).
* Pregnancy or lactation.
* History of seizures.
* Current or past history of asthma and/or the occasional or daily use of albuterol or other beta-agonist inhalers.
* Current use of medications that might affect heart rate or skin conductance.
* Use of carbamazepine or nitroglycerin (or any other medication deemed to be hazardous if taken with NAC) within 14 days of study.
* History of significant hepatic, renal, endocrine, cardiac (i.e., arrhythmia requiring medication, angina pectoris, myocardial infarction,), stroke, seizure, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, metabolic, or other disorders that may place the participant at increased risk per the judgment of the study physician.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were recruited over 9 months in 2008-2009.
Pre-assignment Details: After informed consent, an assessment/screening visit was used to determine if prospective participants met criteria for inclusion. Briefly, participants were required to be regular cannabis users meeting current criteria for dependence. Participants with unstable psychiatric or medical issues were excluded.
Groups:
- N-acetylcysteine: All participants received N-Acetylcysteine 1200 mg twice daily during four weeks of participation. Tolerability, marijuana use, and reactivity to marijuana cues were investigated.
Period: Overall Study
Arm/Group | N-acetylcysteine
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (0.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment, Measured by Number of Participants Recruited and Retained During Study Period
Description: Feasibility of recruiting and retaining participants during the study period. This is the primary outcome of interest for this proof-of-concept feasibility preliminary study.
Time Frame: one year
Measure: Number; unit: Participants
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: Four weeks (full course of treatment)
Arm/Group | N-acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=24)
All (Investigations) | 15 (32)

LIMITATIONS AND CAVEATS:
This was a small, open-label, non-controlled trial, with the associated limitations. A controlled trial is needed to test the effects of N-acetylcysteine relative to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No